CLINICAL TRIAL: NCT05249686
Title: Effects of Two Different Physical Therapy Protocols After an Endodontic Intervention: A Randomized Controlled Trial
Brief Title: Effects of Two Different Physical Therapy Protocols After an Endodontic Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Zaragoza (Other)
Responsible Party: Principal Investigator, Isabel Albarova-Corral, Associate Lecturer in Physiotherapy, Universidad de Zaragoza
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PI18/370
Record Dates: First submitted 2022-02-08; First posted 2022-02-22 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Root Canal Therapy; Endodontically Treated Teeth
Keywords: Dry Needling; Manual Therapy; Temporomandibular Joint; Cervical spine; Root Canal Therapy
MeSH Terms: conditions — Tooth, Nonvital | interventions — Musculoskeletal Manipulations; Dry Needling

STUDY DESIGN:
Intervention Model Description: This will be a randomized controlled trial with 3 different groups
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Manual Therapy + Dry Needling (Experimental)
  Interventions: Other: Manual Therapy + Dry Needling
- Manual Therapy (Active Comparator)
  Interventions: Other: Manual Therapy
- Control (No Intervention): The control group received only the dentist´s usual advice after endodontic surgery.

INTERVENTIONS:
Other: Manual Therapy + Dry Needling — Dry Needling: This is a minimally invasive procedure where a fine needle or acupuncture needle is inserted into the skin and muscle in order to stimulate myofascial trigger points (MTrP) provoking one to six local twitch responses (LTR).
  Manual Therapy Protocol: Intraoral manual techniques were applied to the musculature of both sides, both masseter and medial pterygoid, consisting of both massage and stretching. Furthermore, a grade I-II in the slack-zone traction was applied in the temporomandibular joint (TMJ).
  Arms: Manual Therapy + Dry Needling
Other: Manual Therapy — Manual Therapy Protocol: Intraoral manual techniques were applied to the musculature of both sides, both masseter and medial pterygoid, consisting of both massage and stretching. Furthermore, a grade I-II in the slack-zone traction was applied in the temporomandibular joint (TMJ).
  Arms: Manual Therapy

SUMMARY:
The purpose of this study was to evaluate the clinical results produced by a manual therapy treatment combined with dry needling (MT+DN) and a manual therapy treatment (TM) versus a control (C), to normalize the altered cervico-mandibular variables after a session of root canal therapy.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years old and requiring an endodontic intervention.

Exclusion Criteria:

* Have received TMJ or cervical treatment during the last month, presented any red flag, neurological or cognitive impairment (inability to understand the questionnaires or examination).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2022-03-07 (Actual); Primary Completion 2022-05-07 (Actual); Study Completion 2022-06-07 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline in Maximum Active Mouth Opening at 1 week | Baseline and 1 week
  An electronic caliper (HIBOK DC-516) will be used to measure maximum active mouth opening in supine position. Patients will be instructed to open the mouth as wide as possible without feeling any pain and the distance between upper-lower central incisors (intercisal distance) will be measured in mm.

SECONDARY OUTCOMES:
Mean change from baseline in Pain intensity at 1 week | Baseline and 1 week
  Pain intensity will be measured using a visual analogue scale (VAS) from 0 to 10 (where 0 is no pain and 10 is the worst pain imaginable).
Mean change from baseline in Pressure Pain Threshold (PPT) at 1 week | Baseline and 1 week
  The examiners assess the PPT using a handheld algometer (Wagner, Model FPK). The PPT will be measured bilaterally in the following points of the craniofacial and cervical region: masseter, temporalis, upper trapezius, splenius capitis and suboccipital muscles, and temporomandibular joint. The thenar eminence will be also measured in order to evaluate central sensitization (general pain hypersensitivity) within an intervention-free anatomical location.
Mean change from baseline in Myofascial Trigger Points (MTrPs) at 1 week | Baseline and 1 week
  The following muscles of the temporomandibular and cervical regions will be examined: masseter, temporalis, sternocleidomastoid, upper trapezius, splenius capitis and suboccipital muscles.
Mean change from baseline in Cervical Spine Range of Movement (ROM) at 1 week | Baseline and 1 week
  The examiners assess the cervical ROM using the Clinometer App (version 2.4) for smartphone and a standard goniometer. Cervical flexion, extension, right/left sidebending, right/left rotation, as well as upper cervical spine flexion and extension will be evaluated.
Mean change from baseline in TMD-Pain Screener (TMJ Function) at 1 week | Baseline and 1 week
  The examiners assess temporomandibular disorders (TMDs) using this screening instrument f
Mean change from baseline in Helkimo Index (TMJ Function) at 1 week | Baseline and 1 week
  The examiners assess the severity and pain of TMDs patients using the Helkimo Index.
Mean change from baseline in Jaw Functional Limitation Scale (JFLS-20) (TMJ Function) | Baseline and 1 week
  The examiners assess the functional limitation globally during the last month using the JFLS-20. Subjects must indicate the level of limitation during the last week in a range from 0 to 10.
Mean change from baseline in Neck Disability Index (NDI) (Neck Function) at 1 week | Baseline and 1 week
  The examiners assess the self-perceived disability from neck pain using the NDI.
Mean change from baseline in Headache Impact Test (HIT-6) (Headache Disfunction) at 1 week | Baseline and 1 week
  The examiners assess the impact of headache on patients' lives using the HIT-6.

CONTACTS AND LOCATIONS:
Locations (1):
- Servicio de Prácticas Odontológicas del Grado en Odontología de la Universidad de Zaragoza, Huesca, Aragon, Spain

IPD SHARING:
Plan to Share IPD: No